CLINICAL TRIAL: NCT05603351
Title: ProstaPilot: Prostate Cancer Screening Using MRI With an Abbreviated Protocol
Brief Title: Prostate Cancer Screening With Abbreviated MRI Protocol
Acronym: ProstaPilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk Memorial Cancer Institute (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NU22-09-00539
Record Dates: First submitted 2022-09-02; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: magnetic resonance imaging; biparametric MRI; prostate cancer; PI-RADS; PSA; preventive medicine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging; Biopsy

STUDY DESIGN:
Intervention Model Description: A prospective cross-sectional (with a longitudinal component, 2nd screening round) study evaluating the possibility of using the abbreviated bpMRI protocol technique for screening clinically significant prostate cancer in men from the general population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preventive prostate examination by bpMRI (Experimental): The cohort consists of patients:
  * with age 50-69 years
  * without any contraindications to MRI or biopsy
  * without known status of prostate cancer or prostate biopsy in the past (interventions for BPH are not a restriction)
  * without known BRCA mutation
  * without PSA test or prostate MRI in the past 2 years
  * without any signs of prostatitis or urinary tract infection in the past 6 months.
  Interventions: Diagnostic Test: magnetic resonance; Diagnostic Test: serum PSA examination; Procedure: Biopsy

INTERVENTIONS:
Diagnostic Test: magnetic resonance — biparametric MRI with protocol including anatomical T2 sequence and diffusion-weighted images (DWI), according to the standards
  Other Names: MRI
Diagnostic Test: serum PSA examination — testing of prostate-specific antigen (PSA) in serum
Procedure: Biopsy — Men with a positive MR test are planned for a targeted MRI/US fusion and systematic prostate biopsy.
  Men with a positive blood marker (either PSA, PSAD, or PHI) are planned for a systematic 12 core biopsy. Positive test results are PSA ≥ 3, integrated marker PSAD ≥ 0.15, and PHI ≥ 35.

SUMMARY:
Prostate cancer is one of the most common malignancies in the male population with incidence and mortality rates comparable to breast cancer in women, but in contrast, a population screening program that would fulfill all the recommended criteria is not yet available. According to international recommendations, the preventive PSA sampling used in clinical practice is not suitable because of the concurrent detection of clinically insignificant carcinomas in a major proportion of tests. These clinically non-significant cancers make up a significant and increasing proportion with age. Detection of non-significant cancers burdens the health care system and patients with the care that has no positive impact on their health. Current preventive serum prostate-specific antigen (PSA) testing does not distinguish benign hyperplasia and nonsignificant carcinoma from clinically significant cancer. It is therefore not suitable for full-scale screening.

According to current guidelines, magnetic resonance imaging (MRI) is indicated only in patients with an increased risk of cancer for detection or staging after biopsy and is not used for screening. According to recent studies, MRI has detected an increased proportion of significant cancers in the general population compared to screening based on PSA, while fewer clinically insignificant cancers have been detected. In screening, a shorter examination protocol without contrast medium (biparametric MRI) is used with a lower cost per examination, allowing to increase both the number of patients examined and patient comfort.

The main objective of the project is to assess the contribution of imaging in the screening of clinically significant prostate cancer and to validate the published results in the Czech population, and extend the screening model by the second round of examinations and additional laboratory markers. The secondary aim is to design a subsequent study with a larger number of participants allowing statistical evaluation, similar to the successful breast cancer screening.

DETAILED DESCRIPTION:
A prospective cross-sectional (with a longitudinal component, 2nd screening round) study evaluating the possibility of using the biparametric MRI protocol technique for screening clinically significant prostate cancer in men from the general population.

Tests performed:

* Serum PSA
* PHI calculation (Prostate Health Index) to be performed only if the PSA values are in the range of 2-10 ng/l
* MRI of the prostate (abbreviated biparametric protocol)
* Digital rectal examination (DRE) as part of a clinical visit at a urologist in patients with a positive PSA test
* Biopsy - if indicated

MRI specifications:

* Protocol with anatomical T2 sequence and diffusion-weighted images (DWI), according to the standards
* Typical complete examination time does not exceed 20 minutes, planned acquisition time less than 15 minutes.
* No contrast agent or spasmolytics is injected.

Blinding:

* Every test evaluator (radiologist/urologist) does not know the results of other tests. · MRI reports entered in the registry obligatorily before the biopsy.
* The patient is not informed which test was positive and resulted in an indication for biopsy.
* The pathologist does not know the results of MRI or laboratory tests.

The sequence of tests:

The MRI is assessed with the PI-RADS 2.1 system, each finding is reported on a scale of 1-5. To minimize the detection of non-significant cancers and to reduce the number of biopsies according to the results of the IP1-Prostagram study, a PI-RADS value of 4-5 was chosen as a positive test representation.

Consensual double reading by 2 experienced uroradiologists (at least 400 MRI of the prostate read by the beginning of the study). Men with a positive MRI test are planned for a targeted MRI/US fusion and systematic prostate biopsy.

Men with a positive blood marker (either PSA, PSAD, or PHI) are planned for a systematic 12 core biopsy. Positive test results are PSA ≥ 3, integrated marker PSAD ≥ 0.15, and PHI ≥ 35.

Study participants are invited to repeat the screening tests after 2 years by letter. If they do not respond to a written offer, also by e-mail and SMS.

Definition of clinically significant cancer: • ISUP Grade Group ≥ 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-69 years
* Life expectancy over 10 years
* Ability to undergo all planned procedures (without contraindications to MRI or biopsy)
* No known prostate cancer or prostate biopsy in the past (interventions for BPH are not a restriction)
* No PSA test or prostate MRI in the past 2 years.
* No signs of prostatitis or urinary tract infection in the past 6 months.
* Signed informed consent.

Exclusion Criteria:

* Contraindications to MRI
* Hip replacement
* Known BRCA1/BRCA2 mutation

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the nature of examined organ (prostate), this study is focused exclusively on men.
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the importance of the imaging test in the screening of significant prostate cancer in asymptomatic men, compared with PSA screening: Proportion of positive MRI findings | 2 years
  Proportion of positive MRI findings (PI-RADS 4+) in the general population of men aged 50-69 years.
Distribution of PI-RADS scores in the observed cohort. | 2 years
  Distribution of PI-RADS scores (proportion of individual scores 1-5) in the screened population.
Proportion of positive PI-RADS detections in the cohort of patients indicated for biopsy. | 2 years
  Ratio of significant and non-significant cancers in individual categories of PI-RADS scores in patients indicated for biopsy.

SECONDARY OUTCOMES:
Feasibility evaluation of a larger-scale study of screening for significant prostate cancer using an imaging modality: | 2 years
  Concordance rate (%) between radiologists performing MRI scoring.
Evaluation of complications after an interventional procedure (biopsy). | 2 years
  Number of complications after biopsy.
Evaluation of patient adherence to preventive examination - active recruitment. | 2 years
  Number of participants who agreed to be included in the study through used recruitment strategies.
Patient adherence to preventive examination - self-recruitment. | 2 years
  Number of participants who contacted the team themselves with a request for testing.
Patient adherence to preventive examination. | 2 years
  Number of participants who signed the informed consent and were enrolled in the study.
Evaluation of patient adherence to preventive examination. | 2 years
  Number of participants who visited a screening facility.
Evaluation of patient adherence to preventive examination - completation of planned exams. | 2 years
  Number of participants who completed the designated examination.
Evaluation of the financial burden of the study for the future preventive program of prostate cancer screening. | 2 years
  Costs of individual inclusion and screening tests.
Detection and assessment of potential barriers to patient participation in the study. Assessment of patient adherence to remain in the study throughout the study period. | 2 years
  Numbers and reasons of participants who did not complete scheduled tests, follow-up examinations, or withdrew informed consent.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Staník, MD,PhD., Principal Investigator — Masaryk Memorial Cancer Institute
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loeb S, Bjurlin MA, Nicholson J, Tammela TL, Penson DF, Carter HB, Carroll P, Etzioni R. Overdiagnosis and overtreatment of prostate cancer. Eur Urol. 2014 Jun;65(6):1046-55. doi: 10.1016/j.eururo.2013.12.062. Epub 2014 Jan 9. PMID 24439788
- [Background] Thompson IM, Pauler DK, Goodman PJ, Tangen CM, Lucia MS, Parnes HL, Minasian LM, Ford LG, Lippman SM, Crawford ED, Crowley JJ, Coltman CA Jr. Prevalence of prostate cancer among men with a prostate-specific antigen level < or =4.0 ng per milliliter. N Engl J Med. 2004 May 27;350(22):2239-46. doi: 10.1056/NEJMoa031918. PMID 15163773
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Hugosson J, Roobol MJ, Mansson M, Tammela TLJ, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Carlsson SV, Talala KM, Lilja H, Denis LJ, Recker F, Paez A, Puliti D, Villers A, Rebillard X, Kilpelainen TP, Stenman UH, Godtman RA, Stinesen Kollberg K, Moss SM, Kujala P, Taari K, Huber A, van der Kwast T, Heijnsdijk EA, Bangma C, De Koning HJ, Schroder FH, Auvinen A; ERSPC investigators. A 16-yr Follow-up of the European Randomized study of Screening for Prostate Cancer. Eur Urol. 2019 Jul;76(1):43-51. doi: 10.1016/j.eururo.2019.02.009. Epub 2019 Feb 26. PMID 30824296
- [Background] Draisma G, Boer R, Otto SJ, van der Cruijsen IW, Damhuis RA, Schroder FH, de Koning HJ. Lead times and overdetection due to prostate-specific antigen screening: estimates from the European Randomized Study of Screening for Prostate Cancer. J Natl Cancer Inst. 2003 Jun 18;95(12):868-78. doi: 10.1093/jnci/95.12.868. PMID 12813170
- [Background] Nam RK, Wallis CJ, Stojcic-Bendavid J, Milot L, Sherman C, Sugar L, Haider MA. A Pilot Study to Evaluate the Role of Magnetic Resonance Imaging for Prostate Cancer Screening in the General Population. J Urol. 2016 Aug;196(2):361-6. doi: 10.1016/j.juro.2016.01.114. Epub 2016 Feb 13. PMID 26880413
- [Background] Eldred-Evans D, Burak P, Connor MJ, Day E, Evans M, Fiorentino F, Gammon M, Hosking-Jervis F, Klimowska-Nassar N, McGuire W, Padhani AR, Prevost AT, Price D, Sokhi H, Tam H, Winkler M, Ahmed HU. Population-Based Prostate Cancer Screening With Magnetic Resonance Imaging or Ultrasonography: The IP1-PROSTAGRAM Study. JAMA Oncol. 2021 Mar 1;7(3):395-402. doi: 10.1001/jamaoncol.2020.7456. PMID 33570542
- [Background] van der Leest M, Israel B, Cornel EB, Zamecnik P, Schoots IG, van der Lelij H, Padhani AR, Rovers M, van Oort I, Sedelaar M, Hulsbergen-van de Kaa C, Hannink G, Veltman J, Barentsz J. High Diagnostic Performance of Short Magnetic Resonance Imaging Protocols for Prostate Cancer Detection in Biopsy-naive Men: The Next Step in Magnetic Resonance Imaging Accessibility. Eur Urol. 2019 Nov;76(5):574-581. doi: 10.1016/j.eururo.2019.05.029. Epub 2019 Jun 2. PMID 31167748
- [Background] Drost FH, Osses D, Nieboer D, Bangma CH, Steyerberg EW, Roobol MJ, Schoots IG. Prostate Magnetic Resonance Imaging, with or Without Magnetic Resonance Imaging-targeted Biopsy, and Systematic Biopsy for Detecting Prostate Cancer: A Cochrane Systematic Review and Meta-analysis. Eur Urol. 2020 Jan;77(1):78-94. doi: 10.1016/j.eururo.2019.06.023. Epub 2019 Jul 18. PMID 31326219
- [Background] Schoots IG, Padhani AR, Rouviere O, Barentsz JO, Richenberg J. Analysis of Magnetic Resonance Imaging-directed Biopsy Strategies for Changing the Paradigm of Prostate Cancer Diagnosis. Eur Urol Oncol. 2020 Feb;3(1):32-41. doi: 10.1016/j.euo.2019.10.001. Epub 2019 Nov 7. PMID 31706946
- [Background] Chiu PK, Ng CF, Semjonow A, Zhu Y, Vincendeau S, Houlgatte A, Lazzeri M, Guazzoni G, Stephan C, Haese A, Bruijne I, Teoh JY, Leung CH, Casale P, Chiang CH, Tan LG, Chiong E, Huang CY, Wu HC, Nieboer D, Ye DW, Bangma CH, Roobol MJ. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol. 2019 Apr;75(4):558-561. doi: 10.1016/j.eururo.2018.10.047. Epub 2018 Nov 2. PMID 30396635
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] de Rooij M, Israel B, Tummers M, Ahmed HU, Barrett T, Giganti F, Hamm B, Logager V, Padhani A, Panebianco V, Puech P, Richenberg J, Rouviere O, Salomon G, Schoots I, Veltman J, Villeirs G, Walz J, Barentsz JO. ESUR/ESUI consensus statements on multi-parametric MRI for the detection of clinically significant prostate cancer: quality requirements for image acquisition, interpretation and radiologists' training. Eur Radiol. 2020 Oct;30(10):5404-5416. doi: 10.1007/s00330-020-06929-z. Epub 2020 May 19. PMID 32424596
- [Background] Boesen L, Norgaard N, Logager V, Balslev I, Bisbjerg R, Thestrup KC, Jakobsen H, Thomsen HS. Prebiopsy Biparametric Magnetic Resonance Imaging Combined with Prostate-specific Antigen Density in Detecting and Ruling out Gleason 7-10 Prostate Cancer in Biopsy-naive Men. Eur Urol Oncol. 2019 May;2(3):311-319. doi: 10.1016/j.euo.2018.09.001. Epub 2018 Sep 27. PMID 31200846
- [Background] Eldred-Evans D, Tam H, Sokhi H, Padhani AR, Winkler M, Ahmed HU. Rethinking prostate cancer screening: could MRI be an alternative screening test? Nat Rev Urol. 2020 Sep;17(9):526-539. doi: 10.1038/s41585-020-0356-2. Epub 2020 Jul 21. PMID 32694594
- [Derived] Svetlak M, Standara M, Malatincova T, Stanik M, Miklanek D, Hejcmanova K, Pacal M, Hrabec R, Ngo O, Hejduk K, Kristek J, Uher M, Majek O, Poprach A. Exploring motivations and barriers in prostate cancer screening: lessons from a volunteer-based MRI screening study. Front Public Health. 2025 Nov 17;13:1646494. doi: 10.3389/fpubh.2025.1646494. eCollection 2025. PMID 41334411
- See also: Prostate cancer epidemiology in the Czech republic. — https://www.uroweb.cz/index.php?pg=odborne-analyzy-a-publikace--epidemiologie-nadoru-urogenitalniho-systemu-v-ceske-republice
- See also: Epidemiology of malignant tumors in the Czech republic — https://www.svod.cz

DOCUMENTS (2):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT05603351/Prot_000.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT05603351/ICF_001.pdf